CLINICAL TRIAL: NCT07126054
Title: The Effect of Bibliotherapy Administered During the Preoperative Period on Vital Signs, Anxiety, and Coping With Illness in Adolescent Patients
Acronym: Bibliotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, pınar dogan, Asst.Prof., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 98127364
Record Dates: First submitted 2025-08-09; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Psycho-educational; Anxiety; Illness, Critical
Keywords: Adolescent patient; perioperative period; bibliotherapy; coping with illness; anxiety
MeSH Terms: conditions — Anxiety Disorders; Critical Illness | interventions — Bibliotherapy

STUDY DESIGN:
Intervention Model Description: a pretest-posttest randomized controlled experimental design
Who Masked: Participant
Masking Description: Participant masking indicates a patient with a diagnosis of chronic renal failure receiving hemodialysis treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): As part of the bibliotherapy intervention, the book "My Surgery Journey" (bibliotherapy), developed by the researchers, was read to the patients during in two hours the preoperative period and discussed individually with them, aiming to help the patients understand the surgical process and reduce their anxiety.
  Interventions: Behavioral: bibliotherapy
- Control group (No Intervention): Only routine nursing care and information were continued in this group.

INTERVENTIONS:
Behavioral: bibliotherapy — Bibliotherapy is a therapeutic approach that uses carefully prepared reading materials (My Surgery Story) to support individuals' understanding, coping, and anxiety, facilitated through guided reading and discussion.
  Arms: Intervention group

SUMMARY:
This study aimed to evaluate the effects of bibliotherapy administered to adolescent patients in the preoperative period on vital signs, anxiety levels, and coping attitudes using a pretest-posttest controlled experimental design. The main hypotheses:

H1: Bibliotherapy administered to adolescent patients during the preoperative period positively affects at least one of the patients' vital signs.

H2: Bibliotherapy administered to adolescent patients during the preoperative period reduces the patients' state anxiety level.

H3: Bibliotherapy administered to adolescent patients during the preoperative period reduces the patients' trait anxiety level.

H4: Bibliotherapy administered to adolescent patients during the preoperative period increases the patients' level of coping with illness.

Researchers will compare control group to see if vital signs, anxiety and coping with illnes levels. Bibliotherapy was applied to the intervention group, while the control group received routine clinical care.

DETAILED DESCRIPTION:
The study was conducted with 90 adolescent patients scheduled for surgical intervention at the pediatric surgery clinic of a city hospital. Data were collected using the "Personal Information Form," "Vital Signs Monitoring Form," "State-Trait Anxiety Inventory for Children," and the "Coping Attitudes Assessment Scale. In the intervention group, a three-stage process (pre-test, bibliotherapy, and post-test) was implemented; as part of bibliotherapy, the book "My Surgery Journey" was read to the patients and discussed individually to help them understand the surgical process and reduce anxiety. In the control group, only pre-test and post-test measurements were conducted at the same time intervals, without any psychoeducational intervention. In both groups, vital signs, anxiety levels, and coping with illness were assessed using standardized scales and measurement methods.

ELIGIBILITY:
Inclusion Criteria:

* who were between 10 and 17 years old,
* literate (able to read and write),
* diagnosed with appendicitis and scheduled for surgery,
* without any prior major surgical interventions,
* who, along with their parents, consented to participate in the study.

Exclusion Criteria:

* Failure of the patient to recover physiologically on the 1st and 2nd postoperative days
* Presence of postoperative complications
* Early discharge from the clinic

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Vital sign: pulse | Day 1: Before two hours from surgery and at after eigth hours from surgery (Day 1)
  Pulse is the rhythmic expansion of an artery caused by the ejection of blood from the heart, reflecting the heart rate and rhythm.
Vital sign: blood pressure | Day 1: Before two hours from surgery and at after eigth hours from surgery (Day 1)
  Blood pressure is the force exerted by circulating blood against the walls of the arteries, indicating the pressure during heartbeats (systolic) and between beats (diastolic).
  Ask ChatGPT Blood pressure is the force exerted by circulating blood against the walls of the arteries, indicating the pressure during heartbeats (systolic) and between beats (diastolic).
  Ask ChatGPT Blood pressure is the force exerted by circulating blood against the walls of the arteries, indicating the pressure during heartbeats (systolic) and between beats (diastolic).
vital sign: body temperature | Day 1: Before two hours from surgery and at after eigth hours from surgery (Day 1)
  Body temperature is the measure of the body's ability to generate and dissipate heat, reflecting the balance between heat production and heat loss.
vital sign: respiratory rate | Day 1: Before two hours from surgery and at after eigth hours from surgery (Day 1)
  Breathing, or respiratory rate, is the number of breaths taken per minute, indicating how effectively the body is exchanging oxygen and carbon dioxide.
vital sign: Oxygen saturation | Day 1: Before two hours from surgery and at after eigth hours from surgery (Day 1)
  Oxygen saturation is the percentage of hemoglobin in the blood that is saturated with oxygen, indicating how efficiently oxygen is being transported to body tissues.
State-Trait Anxiety Inventory for Children | Day 1: 1 hour after the decision for surgery is explained to the patient and and at after eigth hours from surgery (Day 1)
  The State-Trait Anxiety Inventory for Children measures both the temporary (state) and general (trait) levels of anxiety experienced by children. The highest possible score on the State Anxiety Inventory is 60, and the lowest is 20. An increase in the score indicates a higher level of anxiety.
Coping Attitudes Assessment Scale | Day 1: 1 hour after the decision for surgery is explained to the patient and and at after eigth hours from surgery (Day 1)
  The Coping Attitudes Assessment Scale evaluates an individual's strategies and attitudes toward managing stress and adapting to challenging situations. The highest possible score on the scale is 160, and the lowest is 40. A higher score on the scale indicates a higher level of coping attitude.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University Hospital, Istanbul, Bağcılar
  - Istanbul Medipol University, Istanbul

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study, including de-identified demographic information, clinical measurements (vital signs), anxiety scores, and coping assessment results, will be made available to other qualified researchers upon reasonable request. All shared data will be fully anonymized to protect participant confidentiality. Data will be accessible starting from [12 months] after publication of the primary results, through a secure data repository or via direct request to the corresponding author. Researchers requesting access will be required to submit a brief proposal outlining the purpose of the data use and agree to data use agreements ensuring ethical and secure handling of the information.